CLINICAL TRIAL: NCT03100448
Title: An Open, Prospective, Multi-center Study Evaluating the On1 Concept on NobelActive Implants
Brief Title: A 1-year Clinical Investigation on the On1 Concept
Acronym: T-190
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-190
Record Dates: First submitted 2017-02-28; First posted 2017-04-04 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2019-10

CONDITIONS: Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- On1 Concept (Other): On1 Concept & NobelActive implants
  Interventions: Device: On1 Concept

INTERVENTIONS:
Device: On1 Concept — NobelActive implant placement with simultaneous On1 Base placement

SUMMARY:
A 1-year Clinical Investigation on the On1 Concept.

DETAILED DESCRIPTION:
This open, prospective, multi-center clinical trial evaluates the On1 Concept for the treatment of patients in need for single tooth replacement or 3-unit bridges in the mandible or maxilla.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 18 years of age (or age of consent) and has passed cessation of growth.
* Obtained informed consent from the subject.
* The patient is willing and able to comply with all study related procedures (such as exercising oral hygiene and attending all follow-up procedures).
* The subject shall be healthy and compliant with good oral hygiene.
* Full-mouth bleeding score (FMBS) lower than 25% [10].
* Full-mouth plaque score (FMPI) lower than 20% [11].
* Suitable for implant treatment in the posterior, pre-molar and canine area in the mandible or maxilla.
* The subject shall have a favorable and stable occlusal relationship.
* In need of one or multiple single tooth replacements or 3-unit bridges.
* Healed sites in need for implant placement (i.e. minimum of 6 weeks post extraction).
* The implant sites are free from infection and extraction remnants.
* The subject is suitable for a 1-stage surgical procedure.
* Sufficient amount of buccal and lingual keratinized mucosa.
* The subject has a sufficient amount of bone for placing NobelActive implants with a length of at least 8 mm.
* Primary implant stability as assessed by manual hand testing.

Exclusion Criteria:

* The subject is not able to give her/his informed consent of participating.
* Health conditions, which do not permit the surgical (including anesthesia) or restorative procedure.
* Reason to believe that the treatment might have a negative effect on the subject's overall situation (psychiatric problems), as noted in subject records or in subject history.
* Any disorders in the planned implant area such as previous tumors, chronic bone disease or previous irradiation in the head/neck area.
* Infections in the planned implantation site or adjacent tissue.
* Acute, untreated periodontitis in the planned implantation site or adjacent tissue.
* Any ongoing application of interfering medication (steroid therapy, bisphosphonate, etc.).
* Uncontrolled diabetes, i.e. a subject with diagnosed diabetes that has a history of neglecting doctor's recommendations regarding treatment, food and alcohol intake or A1c level above 8%.
* Alcohol or drug abuse as noted in subject records or in subject history.
* Smoking of >10 cigarettes/day.
* Fresh extraction sites (up to 6 weeks).
* Severe bruxism or other destructive habits.
* Pregnant or lactating women at the time of implant insertion.
* Previous bone augmentation (lateral and/or vertical).
* Soft tissue augmentation less than 2 months before implant placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Marginal bone remodeling | 12 months
  The change in the marginal bone level around the implants from baseline to 12-months of follow-up is measured on paired radiographs.

SECONDARY OUTCOMES:
Soft tissue outcome (soft tissue height) | 12 months
  The change in soft tissue height from baseline to 12-months of follow-up.
Component Survival | 12 months
  Survival rates of implants as well as On1 components and prosthetics.
Component Success | 12 months
  Success of implants as well as On1 components and prosthetics by clinical evaluation calculated in a cumulative success rate life table.
Patient's pain perception (visual analogue score) | 3 months
  The patient's pain perception during the post surgery period is evaluated by the use of a visual analogue score.
Patient's oral health related quality of life (OHIP-14) | 12 months
  The patient's oral health related quality of life is evaluated by the use of the OHIP-14 questionnaire.
Patient's satisfaction with function & esthetics (visual analogue score) | 12 months
  The patient's satisfaction with function & esthetics is evaluated by the use of a visual analogue score.
Ease of use of the On1 Concept (questionnaire) | 12 months
  The ease of use of the On1 Concept is evaluated by the use of a surgeon questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Alina Gologan, DMD, Study Director — Nobel Bioacare
Locations (6):
- Service de Médecine dentaire CHU Sart Tilman, Liège, Belgium
- Studio Odontoiatrico Specialistico, Cattolica, Italy
- Lithuania (3):
  - Dental Clinic Auksteja, Kaunas, LT
  - Dental Clinic Auksteja, Kaunas
  - Vilnius Implantology Center, Vilnius
- Tandartspraktijk Staas & Bergmans, 's-Hertogenbosch, Netherlands

IPD SHARING:
Plan to Share IPD: No